CLINICAL TRIAL: NCT02609373
Title: Improving Cancer-Related Outcomes in Shift Workers
Acronym: ICOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Carolyn Gotay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-701007
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: shiftwork; sleep hygiene; prevention; intervention; occupational; biological; breast cancer; lifestyle
MeSH Terms: conditions — Breast Neoplasms; Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sleep intervention (Other): Sleep intervention
  Interventions: Behavioral: Sleep intervention

INTERVENTIONS:
Behavioral: Sleep intervention — Session 1: Intervener & participant review 2-week sleep diary and actigraph data. Provide individualized sleep hygiene prescription.
  Session 2: Review sleep diary; calculate sleep efficiency; identify adjustments needed.
  Session 3: Review sleep-related vs. stress-related symptoms. Develop plan for sleep-related symptoms and discuss "Sleep Restriction with Relaxation Exercises." Session 4: Reinforce progress and make corrections as required. If Sleep Restriction is not working, Stimulus Control is introduced.
  Session 5-10: Provide reinforcement, assess adherence, answer questions, and offer encouragement and monitoring, including alterations as required.
  Booster sessions: At 8 & 10 months: reinforcement, question answering, encouragement and monitoring.

SUMMARY:
Shift work with circadian disruption has been linked with increased breast cancer incidence. The mechanisms for this effect are not yet completely understood.

This study evaluates the impact of a previously developed sleep intervention in shift workers at risk of breast cancer; and assesses mediating variables that may explain the relationship between shift work and breast cancer.

A sample of women night shift workers were provided with a sleep intervention. The intervention is a standard approach used in a sleep clinic and is delivered by telephone by a trained intervener.

Hypothesis: The intervention will improve sleep in women night shift workers, which will in turn have a positive impact on biological and behavioural risk factors associated with breast cancer and quality of life.

DETAILED DESCRIPTION:
47 female night shift workers completed a sleep intervention. The intervention follows an established sleep therapy protocol. Assessments at baseline, 6 and 12 months include mammographic density and possible mediating variables known to be linked to breast cancer risk including behavioural, biometric, and biological measures. Behavioural and self-report measures of sleep quality and physical activity are assessed as well as self-reported chronotype and quality of life.

The intervention is a multi-session intervention using cognitive behavioural principles to increase healthy sleep by addressing a variety of behaviours that may influence sleep quality and quantity, based an established telephone-based protocol used at the UBC Hospital Sleep Disorders Clinic. It includes 10 telephone sessions spaced over a 6-month period, and 2 additional booster sessions at 8 and 10 months. Participants are given a sleep diary at baseline to complete for 2 weeks before the sleep hygiene telephone counseling session begins.

The intervention protocol incorporates sleep assessment, maintaining a sleep diary and use of an actiwatch (to measure sleep and physical activity), sleep hygiene (i.e., controlling behavioural and environmental factors that affect sleep), stimulus control therapy (i.e., teaching individuals how to eliminate behaviours that are incompatible with sleep), sleep restriction therapy (i.e., teaching how to limit time in bed to time asleep), cognitive restructuring (i.e., modifying non-adaptive thoughts and triggers for insomnia), and relapse prevention. The structured counseling protocol includes concrete exercises and activities, questions and answers, and problem solving strategies.

Medication use is not part of this protocol; if participants wish to explore pharmacologic approaches, they are advised to consult with their physicians. Although some shift workers have received care from the Sleep Clinic in the past, there has not been a systematic focus on this group.

The project manager conducts a telephone-based evaluation of the intervention 6 months post-sleep intervention. Blood and salivary samples are collected using standardized data collection methods at baseline, 6, and 12 months, and mammographic films are collected at baseline and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-65 years
* Working or living in Greater Vancouver Area
* Read and understand English
* Work rotating or permanent night shift at least 3 times per month, for at least 2 years
* Received a screening mammogram within the past 3 years

Exclusion Criteria:

* History of breast cancer
* On active cancer therapy for any cancer
* Pregnant
* Diabetes requiring drug treatment

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality | Baseline, 6 months
  Self-reported "good" sleep quality at baseline and 6 months

SECONDARY OUTCOMES:
Change in melatonin | Baseline, 6 months
  Change in melatonin at baseline and 6 months
Change in melatonin | 6 months, 12 months
  Change in melatonin at 6 and 12 months
Change in melatonin | Baseline, 12 months
  Change in melatonin at baseline and 12 months
Change in cortisol | Baseline, 6 months
  Change in cortisol at baseline and 6 months
Change in cortisol | 6 months, 12 months
  Change in cortisol at 6 and 12 months
Change in cortisol | Baseline, 12 months
  Change in cortisol at baseline and 12 months
Change in breast density | Baseline, 12 months
  Change in breast density at baseline and 12 months
Change in IGF-1 and IGFBP 1,2,3,7 | Baseline, 6 months
  Change in IGF-1 and IGFBP 1,2,3,7 at baseline and 6 months
Change in IGF-1 and IGFBP 1,2,3,7 | 6 months,12 months
  Change in IGF-1 and IGFBP 1,2,3,7 at 6 and 12 months
Change in IGF-1 and IGFBP 1,2,3,7 | Baseline, 12 months
  Change in IGF-1 and IGFBP 1,2,3,7 at baseline and 12 months
Change in Vitamin D | Baseline, 6 months
  Change in Vitamin D at baseline and 6 months
Change in Vitamin D | 6 months, 12 months
  Change in Vitamin D at 6 and 12 months
Change in Vitamin D | Baseline, 12 months
  Change in Vitamin D at baseline and 12 months
Change in C-reactive protein | Baseline, 6 months
  Change in C-reactive protein from baseline to 6 months
Change in C-reactive protein | 6 months and 12 months
  Change in C-reactive protein from 6 to 12 months
Change in C-reactive protein | Baseline, 12 months
  Change in C-reactive protein from baseline to 12 months
Change in insulin | Baseline, 6 months
  Change in insulin from baseline to 6 months
Change in insulin | 6 months and 12 months
  Change in insulin from 6 to 12 months
Change in insulin | Baseline, 12 months
  Change in insulin from baseline to 12 months
Change in glucose | Baseline, 6 months
  Change in glucose from baseline to 6 months
Change in glucose | 6 months and 12 months
  Change in glucose from 6 to 12 months
Change in glucose | Baseline, 12 months
  Change in glucose from baseline to 12 months
Change in quality of life | Baseline, 6 months
  Change in quality of life from baseline to 6 months
Change in quality of life | 6 months, 12 months
  Change in quality of life from 6 months to 12 months
Change in quality of life | Baseline,12 months
  Change in quality of life from baseline to 12 months
Intervention Evaluation | 12 months
  Participant satisfaction and perceptions of intervention assessed by semi-structured telephone interview
Change in sleep quality | 6 months, 12 months
  Self-reported "good" sleep quality at 6 and 12 months
Change in sleep quality | Baseline, 12 months
  Self-reported "good" sleep quality at baseline and 12 months
Change in health and lifestyle | Baseline, 6 months
  Change in self-reported health and lifestyle assessed by structured questionnaire at baseline and 6 months
Change in health and lifestyle | 6 months, 12 months
  Change in self-reported health and lifestyle assessed by structured questionnaire at 6 and 12 months
Change in health and lifestyle | Baseline, 12 months
  Change in self-reported health and lifestyle assessed by structured questionnaire at baseline and 12 months

OTHER OUTCOMES:
Concordance between self-reported sleep quality and other indicators | Baseline, 6 months, 12 months
  Comparison of ratings between self-reports, diary data, and actigraph readings at all time points

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Gotay, PhD., Principal Investigator — The Univeristy of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No